CLINICAL TRIAL: NCT00179413
Title: Phase IV Study of Long Term Peg-Intron for Patients Who Have Failed to Respond to Rebetron/Interferon With Advanced Fibrosis and Cirrhosis Secondary to Hepatitis C- The Copilot Trial
Brief Title: Study of Long-term Peg Intron vs. Colchicine in Non-responders.
Acronym: COPILOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Nezam H. Afdhal, Professor of Medicine, Part-time, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2001P000002
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis C Virus; Advanced Fibrosis; Cirrhosis
Keywords: hepatitis C; cirrhosis; interferon; colchicine
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — peginterferon alfa-2b; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-Intron (Active Comparator): PEG-Intron 0.5mcg/kg once a week SC
  Interventions: Drug: PEG -Intron
- Colchicine (Active Comparator): 0.6mg twice a day
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: PEG -Intron
  Other Names: PEG interferon Alfa-2b 0.5mcg/kg weekly
  Arms: PEG-Intron
Drug: Colchicine — 0.6mg twice a day
  Arms: Colchicine

SUMMARY:
In this study Peg-Intron will be tested to see if it will give better results than Colchicine. At this time, there is currently no recommended maintenance treatment for patients who have failed to respond to Interferon/Rebetron/Peg Intron and have advanced fibrosis. The purpose of this study is to compare two treatments to slow down the progression of liver disease and to prevent liver failure and liver cancer. The treatment will not cure Hepatitis C, but is being evaluated to see if it can slow down disease progression.

DETAILED DESCRIPTION:
We are proposing a randomized trial of Peg-Intron 0.5mcg per kg weekly versus colchicine 0.6mg bid in prior non-responders to Interferon, Rebetron, PegIntron, or PegIntron & Ribavirin or any third agent such as Pegasys, CellCept, Amantadine with advanced fibrosis/cirrhosis. The specific aims of this proposal are to evaluate the role of long term Peg-Intron therapy on the natural history of patients with advanced chronic HCV infection with a primary focus on prevention of hepatic decompensation, progression of fibrosis and hepatoma development.

The study design will focus on 3 monthly clinical evaluation for decompensation of liver function, rigorous clinical screening for development of hepatocellular cancer and liver biopsies for determination of progression of liver fibrosis every second year.

ELIGIBILITY:
Inclusion Criteria:

* *Adult male or female, age 18 to 75 years

  * HCV RNA positive by PCR
  * Previous treatment with at least three months of interferon or interferon / Ribavirin. Patients should have had no interferon for at least 2 months prior to enrollment.

    1. Non-responders are identified by failure to clear virus by PCR after a minimum 3-month course of treatment and who have been off treatment for at least 2 months with a positive PCR for HCV prior to entry into the current study, 2) Partial responders have a reduction of 1 long in HCV RNA, but the virus is still detectable, 3) Breakthrough patients have been negative on treatment, but virus appeared while still on treatment, 4) Relapsers are defined as negative PCR at some point during treatment, but virus reoccurred or was detectable by HCV PCR when treatment stopped.

Patients should have had a liver biopsy showing at least Stage 3 disease prior to being considered for this study. A baseline liver biopsy is necessary for inclusion in the study. Baseline liver biopsies can be performed within six months of entering the study.

In patients with cirrhosis and endoscopic evidence of portal hypertension, a biopsy within the last 2 years is acceptable as the baseline biopsy. For patients with established cirrhosis on liver biopsy and no portal hypertension, a biopsy within 12 months can be used as the baseline biopsy if it is available for evaluation by the Pathology core. All these patients will still require liver biopsy at 2 years and 4 years. The decision to biopsy at 2 and 4 years is also a clinical decision and in the presence of clinical progression or coagulopathy, or where there may be a risk from liver biopsy, the Investigator should call the PI, Dr. Afdhal for a waiver of biopsy. Patients with Ishak Stage 3 and 4 require a biopsy within 6 months of randomization.

* Hemoglobin >= 11 g/dl in males and 10 g/dl in females
* Neutrophil count > 1,500/mm3
* Platelets > 50, 000/mm3

Platelet count: For standard dose of PEG-Intron 0.5mcg/kg platelet count must be greater than 70,000. Patients with platelet count 50 - 70,000 can start at 0.25mcg/kg for weeks 0 - 4. If platelets fall to less than 30,000, stop treatment. If platelets remain > 50,000 at week 4, PEG-Intron can be increased to 0.5mcg/kg. Patients randomized to Colchicine with platelets 50,000 - 70,000 can be started at standard dose 0.6mg bid po with standard dose reduction.

* Prothrombin time <= 3secs prolonged compared to control or an equivalent INR < 1.5
* Total bilirubin < 3gm/dL
* Fasting blood sugar <= 115 mg/dl or within 20% of the upper limit of normal for non-diabetic patients
* Albumin (> 2.8mg/dl)
* Serum creatinine < 1.4 mg/dL
* TSH within the normal range (Patients with thyroid disease who are well controlled are eligible if the remainder of the inclusion/exclusion criteria are met)
* HIV negative.

  * HBsAg negative
  * Childs Pugh score of less than or equal to 7
  * Serum positive for anti-hepatitis C antibodies or HCV RNA.
  * Alpha-fetoprotein < 100ng/ml with ultrasound negative for focal mass or HCC. For any patient with an Alpha-fetoprotein >100 ng/ml either a triple phase contrast CT scan or MRI with gadolinium must show no focal mass or evidence of HCC
  * Ultrasound with no evidence of focal mass suggestive of hepatoma (within 6 months of informed consent).
  * Documentation that sexually active female patients of childbearing potential are practicing adequate contraception during the treatment period. A urine pregnancy test obtained at entry prior to the initiation of treatment must be negative. Female patients must not be breast-feeding. Documentation that sexually active male patients are practicing acceptable methods of contraception during the treatment period.
  * Written informed consent specific for this protocol has been obtained prior to entry.

Exclusion Criteria:

* Any cause of liver disease based on patient history and biopsy (where applicable) other than chronic hepatitis C including but not limited to:

  * Co-infection with hepatitis B or HIV
  * Hemochromatosis (confirmed by genetic testing)
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Renal or liver transplant patients
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Obesity induced liver disease
  * Drug related liver disease

In addition:

* Evidence of decompensated liver disease such as a history or presence of ascites, and spontaneous encephalopathy. Patients with past bleeding esophageal varices that have not bled for more than 1 year can be included.
* Hypersensitivity to alpha interferon
* Drug related liver disease
* Hemoglobinopathies (e.g. Thalassaemia, sickle cell disease).
* Patients with clinically significant retinal abnormalities.
* Substance abuse, such as alcohol (·> 80 gm/day), I.V. drugs and inhaled drugs. If the patient has a history of substance abuse, to be considered for inclusion into the protocol, the patient must have abstained from using the abused substance for at least 6 months. Patients on methadone will be allowed in the study with no restrictions as is now standard of care in HCV therapy.
* Patients with a history of organ transplantation will be excluded.

Preexisting psychiatric conditions, especially depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt are excluded. Patients with a history of mild depression may enter the protocol if they meet the following eligibility criterion and are monitored more intensively.

Mild depression: to include either situational depression of a limited period or depressive symptoms, which do not significantly interfere with the patient's work or daily functions.

Any patient with an active manic element to his/her previous symptom complex will be excluded.

Any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study such as:

* Pre-existing psychiatric condition, especially severe depression, or a history of severe psychiatric disorder
* CNS trauma or seizure disorder requiring therapy
* Significant cardiac dysfunction in the previous 6 months e.g. angina, CCF, hypertension or arrhythmia Patients on treatment are eligible as long as they have been symptom free for the previous 6 months.
* Poorly controlled diabetes mellitus
* Chronic pulmonary disease (e.g. COAD)
* Immunologically mediated diseases (e.g. inflammatory bowel disease, SLE, ITP, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis, severe psoriasis)
* Clinical gout
* Patients with clinically significant retinal abnormalities
* Patients with organ transplants

Any other condition, which in the view of the investigator, would make the patient unsuitable for enrolment, or could interfere with the patient participating in and completing the protocol are included as well.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2000-01-15 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2010-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nezam H Afdhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (49):
- United States (49):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - UAMS Medical Center, Little Rock, Arkansas
  - 34th Street Community Health Center, Bakersfield, California
  - UC Davis Medical Center, Sacramento, California
  - Kaiser Permanende-GI Department, Sacramento, California
  - Gastroenterology Associates, San Diego, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Bruce Stein, MD, Manchester, Connecticut
  - Connecticut Gastroenterology Consultants, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Bach and Godofsky Infectious Disease, Bradenton, Florida
  - Southern Clinical Research Consultants, Hollywood, Florida
  - Gastroenterology Associates of South Florida, South Miami, Florida
  - Digestive Health Services, Downers Grove, Illinois
  - Digestive Disease Associates, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Hampshire Gastroenterology, Florence, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Wayne State University/Haper Hospital, Detroit, Michigan
  - Gastroenterology Division Veterans Affairs Medical Center, Minneapolis, Minnesota
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Gastroenterology Associates, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - VA New Jersey Healthcare System, East Orange, New Jersey
  - Atlantic Gastroenterology, Egg Harbor, New Jersey
  - Florham Park Endoscopy Center, Florham Park, New Jersey
  - Northern New Mexico Gastroenterology, Santa Fe, New Mexico
  - Dr. Sam Moskowitz, MD, PC, Forest Hills, New York
  - Liberty Medical, LLP, New York, New York
  - Metro Medical, New York, New York
  - Columbia University, New York, New York
  - Peter Varunok, MD, Poughkeepsie, New York
  - Upstate Medical Center, Syracuse, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Guthrie Research Foundation, Sayre, Pennsylvania
  - University Gastroenterologists, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Nashville Gastroenterology Specialists Incorporated, Nashville, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - G.I. and Liver Associates, Granbury, Texas
  - Digestive Disease Center, San Antonio, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Health Science Center, Salt Lake City, Utah
  - Medical Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-Intron: PEG-Intron 0.5mcg/kg once a week SC
  PEG -Intron
Period: Overall Study
Arm/Group | PEG-Intron | Colchicine
Started | 282 | 267
Completed | 157 | 152
Not Completed | 125 | 115
Not completed — Adverse Event | 38 | 20
Not completed — Withdrawal by Subject | 87 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-Intron | Colchicine | Total
Number analyzed (Participants) | 282 | 267 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (8.4) | 50.4 (7.1) | 50.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 77 | 167
  Male | 192 | 190 | 382
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 36 | 72
  White | 240 | 227 | 467
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 282 | 267 | 549

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Effect of PEG-Intron 0.5mg Per kg Weekly sc Versus Colchicine 0.6mg Bid Daily on:
Description: number of patients with a liver related outcomes including: mortality, liver transplant, variceal or portal hypertensive bleeding,Development of jaundice, ascites or encephalopathy with an increase in CPT of > 2 points and development of hepatoma
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | PEG-Intron | Colchicine
Number analyzed (Participants) | 282 | 267
Participants | 53 | 59

2. Secondary Outcome: Evaluation of Safety and Tolerability of Long Term Maintenance PEG-Intron in Patients With Cirrhosis
Description: Defined as the number of patients who discontinued therapy due to an adverse event side
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | PEG-Intron | Colchicine
Number analyzed (Participants) | 282 | 267
Participants | 38 | 20

3. Secondary Outcome: Development of Portal Hypertension
Description: Number of patients who develop endoscopic evidence of varices over 4 year period
Time Frame: 4 years
Population: The number of patients at risk include only those patients who at the baseline endoscopy had no evidence of portal hypertension or varices
Measure: Count of Participants; unit: Participants
Arm/Group | PEG-Intron | Colchicine
Number analyzed (Participants) | 92 | 92
Participants | 12 | 24

ADVERSE EVENTS:
Time Frame: Four years on treatment
Description: Although not included as an Adverse event in the clinical trial design but rather as a primary endpoint, liver disease progression has now been added as an adverse event
Arm/Group | PEG-Intron | Colchicine
Serious Adverse Events (participants affected / at risk) | 90/282 | 79/267
Other Adverse Events (participants affected / at risk) | 257/282 | 44/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=282) | Colchicine (N=267)
Depression (Nervous system disorders) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Fatigue, asthenia (General disorders) | 31 (31) | 15 (15)
Disease progression (Hepatobiliary disorders) | 53 (53) | 59 (59) — Patients who met the primary endpoints of disease progression with liver failure, bleeding or liver cancer
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=282) | Colchicine (N=267)
flu like symptoms (General disorders) | 242 (242) | 8 (8)
diarrhea (Gastrointestinal disorders) | 15 (15) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No